CLINICAL TRIAL: NCT07314086
Title: A Clinical Effectiveness Study of Total Laparoscopic Subcutaneous Gland Resection Combined With Nipple-Areola Complex Lift in the Management of Moderate to Severe Gynecomastia in Males
Status: Active, not recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 20251129
Record Dates: First submitted 2025-12-17; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-11

CONDITIONS: Gynecomastia
Keywords: gynecomastia; laparoscopic surgery
MeSH Terms: conditions — Gynecomastia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental group: the group undergoing laparoscopic surgery combined with NAC lift
- control group: the group undergoing simple laparoscopic surgery

SUMMARY:
This study aims to evaluate and compare the treatment outcomes of total laparoscopic subcutaneous gland resection combined with nipple-areola complex (NAC) lift surgery against those of isolated laparoscopic surgery in the management of moderate to severe gynecomastia (GYN) in males.

DETAILED DESCRIPTION:
Gynecomastia (GYN), characterized by unilateral or bilateral breast enlargement, has an incidence ranging from approximately 32.0% to 64.6%, with a progressively increasing trend observed in recent years . Clinically, GYN is categorized into primary and secondary forms: the former is associated with physiological fluctuations in hormonal levels, whereas the latter is primarily attributable to underlying metabolic or neoplastic conditions, as well as medication use. Surgical intervention remains the mainstay of treatment for persistent or symptomatic cases. Given that the male breast is a solid, non-cavitary organ, conventional open surgical approaches have traditionally employed periareolar, crescentic, or double-ring incisions to excise subcutaneous glandular tissue . These techniques, however, are often associated with conspicuous scarring, suboptimal cosmetic results, and relatively high rates of postoperative complications. The advent of liposuction and tumescent lipolysis techniques in the 1990s overcame the technical challenge of cavity creation, thereby facilitating the development of endoscopic approaches. Over the past decade, significant advancements have been achieved through the integration of lipolysis and non-lipolysis techniques, concealed incision sites (e.g., axillary or lateral thoracic approaches), multi-port and single-port endoscopic systems, and robotic-assisted surgery using the Da Vinci Si platform . As a result, the therapeutic objective has evolved from mere glandular excision toward achieving optimal aesthetic outcomes with minimal visible scarring. The 2021 Expert Consensus and Operational Guidelines for Endoscopic Surgery in Breast Diseases established the 5S principles for GYN surgery: (1) complete removal of glandular tissue (sweep); (2) placement of inconspicuous, hidden incisions (scarless); (3) bilateral symmetry; (4) restoration of normal male chest contour (shape); and (5) smooth postoperative skin surface (smoothing) . Nevertheless, in patients with moderate to severe GYN, redundant skin following endoscopic resection frequently leads to malposition of the nipple-areola complex (NAC), including ptosis, depression, or wrinkling, which compromises skin smoothness and undermines both the 5S goals and overall aesthetic satisfaction. To address this limitation, our research team has developed an innovative technique termed the "Nipple-Areola Complex (NAC) Aesthetic Wrinkle-Reducing Band Lifting and Fixation Technique." This minimally invasive approach effectively manages postoperative skin redundancy without additional incisions, enabling precise repositioning of the NAC and improving skin contour. Statistical analysis demonstrates that this technique contributes significantly to enhancing aesthetic outcomes and patient satisfaction in the management of moderate to severe GYN.

ELIGIBILITY:
Inclusion Criteria:

(1) Those with bilateral breast development confirmed by preoperative ultrasound examination; (2) For bilateral developed breasts, the preoperative classification according to Simon's system (hereinafter referred to as Simon classification) is all at grade IIA or above.

Exclusion Criteria:

(1) Benign and malignant tumors of the male breast; (2) Other diseases such as testicular tumors, congenital testicular dysplasia syndrome, hyperthyroidism, liver cirrhosis, primary gonadal hypofunction and oral medications can lead to secondary male breast development; (3) Patients with severe primary diseases such as cardiovascular and cerebrovascular diseases, liver and kidney diseases, and coagulation disorders are not suitable for anesthesia and surgery; (4) Patients with incomplete clinical case data.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe GYN conditions who were treated at the Breast Surgery Department of the First Affiliated Hospital of Harbin Medical University were included.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Differences in the clinical index between the two groups | Baseline
  The patients were divided into two groups: laparoscopic surgery in conjunction with NAC lift group,isolated laparoscopic surgery group. IBM SPSS 27.0 software was used for statistical analysis. The analysis attempt to reveal the differences between the two groups in terms of surgical time, blood loss, and drainage tube placement duration
Difference in the pre- and postoperative convexity of breast between the two groups | Baseline
  The patients were divided into two groups: laparoscopic surgery in conjunction with NAC lift group,isolated laparoscopic surgery group. IBM SPSS 27.0 software was used for statistical analysis. The analysis attempt to reveal the differences between the two groups in terms of the pre- and postoperative convexity of breast
Difference in the recovery rate of skin flatness between the two groups | Baseline
  The patients were divided into two groups: laparoscopic surgery in conjunction with NAC lift group,isolated laparoscopic surgery group. IBM SPSS 27.0 software was used for statistical analysis. The analysis attempt to reveal the differences of the recovery rate of skin flatness between the group undergoing laparoscopic surgery combined with NAC lift and he group undergoing simple laparoscopic surgery at 3, 6, and 12 months postoperatively
Difference in the positioning of the NAC between the two groups | Baseline
  The patients were divided into two groups: laparoscopic surgery in conjunction with NAC lift group,isolated laparoscopic surgery group. IBM SPSS 27.0 software was used for statistical analysis. The analysis attempt to reveal the differences between the two groups in terms of the positioning of the NAC
Differences in the postoperative patient satisfaction between the two groups | Baseline
  The patients were divided into two groups: laparoscopic surgery in conjunction with NAC lift group,isolated laparoscopic surgery group. IBM SPSS 27.0 software was used for statistical analysis. The analysis attempt to reveal the differences between the two groups in terms of postoperative patient satisfaction

SECONDARY OUTCOMES:
Differences in the postoperative complications between the two groups | baseline
  The patients were divided into two groups: laparoscopic surgery in conjunction with NAC lift group,isolated laparoscopic surgery group. IBM SPSS 27.0 software was used for statistical analysis. The analysis attempt to reveal the differences between the two groups in terms of the postoperative complications

CONTACTS AND LOCATIONS:
Locations (1):
- First affiliated hospital of Harbin medical university, Harbin, Heilongjing, China

IPD SHARING:
Plan to Share IPD: No